CLINICAL TRIAL: NCT04549428
Title: Atezolizumab Plus 8 Gy Single-fraction Radiotherapy for Advanced, Oligoprogressive NSCLC After Upfront Chemotherapy and Anti-PD1 Immunotherapy: A Multicentre, Single Arm, Phase II Study
Brief Title: Atezolizumab Plus 8 Gy Single-fraction Radiotherapy for Advanced Oligoprogressive NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for futility, as determined by an interim data analysis.
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Ente Ospedaliero Cantonale, Bellinzona (Other); Istituto Cantonale di Patologia (Other); Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOSI-LUNG-001
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Atezolizumab will be administered at a fixed dose of 1,200 mg by intravenous infusion every 21 days on an outpatient basis until progression, intolerance or loss of clinical benefit, according to the its approved prescribing information. Palliative radiation therapy will be delivered concomitant to the 2nd dose of atezolizumab as a single fraction of 8 Gy
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Intravenous infusion every 21 days, until disease progression, intolerance or loss of clinical benefit.
  Other Names: Tecentriq

SUMMARY:
Multicentre, phase II, open-label, single-arm study evaluating the preliminary efficacy, safety and tolerability of atezolizumab in association with palliative radiotherapy in adult patients diagnosed with advanced (stage IV) NSCLC, irrespective of PD-L1 status, and who have oligoprogressed to both immunotherapy with an anti PD-1 agent (e.g., pembrolizumab or nivolumab) and 1 line of chemotherapy.

DETAILED DESCRIPTION:
Atezolizumab will be administered at a fixed dose of 1,200 mg by intravenous infusion every 21 days on an outpatient basis according to the its approved prescribing information. Palliative radiation therapy will be delivered concomitant to the 2nd dose of atezolizumab as a single fraction of 8 Gy to all eligible metastatic and primary sites.

ELIGIBILITY:
Inclusion Criteria

1. Signed Informed Consent Form
2. Male or female aged ≥ 18 years
3. Ability to comply with the procedures of the study protocol, in the investigator's judgment
4. Histologically or cytologically confirmed diagnosis of metastatic (Stage IV) NSCLC as per the American Joint Committee on Cancer (AJCC) 8th edition
5. No sensitizing EGFR mutation (L858R or exon 19 deletions), ALK fusion oncogene or ROS1 rearrangement detected
6. Progressing to one line of chemotherapy defined as follows:a) A platinum-doublet.

   b) In case of patients being ineligible for platinum-containing regimens but otherwise compliant with the other inclusion-exclusion criteria of the present study, at least one line of mono-chemotherapy is required.

   c) As an exception, patients with oligoprogression to anti PD-1 agents alone for whom the investigator considers local treatment of metastases and continuation of immunotherapy appropriate (i.e. would not be eligible for 2nd line treatment) may be enrolled without a previous line of chemotherapy. In this case, approval by the Project Leader is necessary.
7. Progressing to an anti-PD-1 agent, either associated to chemotherapy or as monotherapy (e.g., pembrolizumab or nivolumab)
8. Life expectancy ≥ 8 weeks
9. Patients with treated, asymptomatic central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria:

   1. Measurable disease outside CNS.
   2. Only supratentorial and cerebellar metastases allowed (i.e., no metastases to midbrain, pons, medulla or spinal cord).
   3. No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed.
   4. No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to initiating study treatment.
   5. No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study.
   6. Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible without the need for an additional brain scan prior to initiating study treatment, if all other criteria are met, including clinical confirmation of no evidence of interim disease progression
10. Measurable disease by RECIST v1.1. Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease.
11. Oligoprogressive disease defined as follows:

    1. A minimum of 1 and a maximum of 4 progressing lesions (with up to 3 total organs and 3 lesions per organ, except skeletal lesions) as assessed by a Positron Emission Tomography-Computed Tomography (PET-CT) scan (contrast enhanced).
    2. Definition of progression is made by RECIST 1.1 criteria (new lesions or increased pre-existing ones).
12. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to initiating study treatment:

    a) Absolute neutrophil count ≥ 1,500 cells/μL without granulocyte colony-stimulating factor support b) White blood cell (WBC) counts > 2,500/μL c) Lymphocyte count > 500/μL d) Serum albumin > 2.5 g/dL e) Platelet count ≥ 100,000/μL without transfusion within 2 weeks of laboratory test used to determine eligibility f) Hemoglobin ≥ 9.0 g/dL, patients may be transfused or receive erythropoietic treatment to meet this criterion g) Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALK) ≤ 2.5 × ULN with the following exceptions: patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN; patients with documented liver or bone metastases: ALK ≤ 5 × ULN.

    h) Serum bilirubin ≤ 1.5 × ULN. Patients with known Gilbert's syndrome who have serum bilirubin level ≤ 3 × ULN may be enrolled i) Serum creatinine ≤ 1.5 × ULN
13. For female patients of childbearing potential agreement to remain abstinent (refrain from heterosexual intercourse) or to use highly effective form(s) of contraceptive methods that result in a failure rate of < 1% per year when used consistently and correctly during the treatment period and for at least 5 months after the last dose of atezolizumab.

    1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
    2. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, and established, proper use of hormonal contraceptives that inhibit ovulation (combined estrogen and progestogen containing hormonal contraception, or progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide), hormone-releasing intrauterine devices, and copper intrauterine devices
    3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
    4. Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drug.
    5. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.

Exclusion criteria

Cancer-specific exclusion criteria

1. Patients with an ECOG Performance status >2
2. Active or untreated CNS metastases as determined by Computed Tomography (CT) or magnetic resonance imaging (MRI) evaluation of the brain during screening and prior radiographic assessments
3. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to initiating study treatment
4. Leptomeningeal disease.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed.
6. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium or >3 mmol/L of corrected serum calcium) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab (patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible; patients who are receiving denosumab to prevent or for mild hypercalcemia prior to enrollment must be willing and eligible to discontinue its use and replace it with a bisphosphonate instead while on study.)
7. History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g. expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, breast ductal carcinoma in situ treated surgically with curative intent).
8. NCI CTCAE Grade 3 or higher toxicities due to any prior therapy (e.g., radiotherapy) (excluding alopecia), which have not shown improvement and are strictly considered to interfere with current study medication, with special focus on prior toxicity to anti-PD1 agents.

General medical exclusion criteria

1. Women who are pregnant or lactating, or intending to become pregnant during the study. Women of childbearing potential including women who have had a tubal ligation, must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.
2. History of autoimmune disease. Exceptions are:

   a) Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible for this study.

   b) Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this study.

   c) Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
   * Rash must cover less than 10% of body surface area (BSA)
   * Disease is well controlled at baseline and only requiring low potency topical steroids
   * No acute exacerbations of underlying condition within the last 12 months requiring treatment with either psoralen plus ultraviolet radiation (PUVA), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors or high potency or oral steroids
3. History of idiopathic pulmonary fibrosis (IPF), organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
4. Known positivity for human immunodeficiency virus (HIV)

   a) Testing is not required in the absence of clinical symptoms and signs suggestive of HIV infection.

   b) Patients with a past history of/or symptoms of HIV are eligible only if serological tests are negative.
5. Known active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or known active hepatitis C a) Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and hepatitis B surface antibody [HBsAb] and absence of HBsAg) are eligible. HBV DNA test must be performed if HBcAb is positive and HBsAb and HBsAg are negative, and in this case, a positive viremia excludes the patient from eligibility. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
6. Severe infections within 4 weeks prior to initiating study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
7. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to initiating study treatment, unstable arrhythmias, or unstable angina.

   a) Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction (LVEF) < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
8. Major surgical procedure other than for diagnosis within 4 weeks prior to initiating study treatment or anticipation of need for a major surgical procedure during the course of the study
9. Prior allogeneic bone marrow transplantation or solid organ transplant
10. Any serious medical condition (including metabolic dysfunction, physical examination finding) or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study or that may affect the interpretation of the results or render the patient at high risk for treatment complications
11. Patients with an illness or condition that may interfere with capacity or compliance with the study protocol, as per investigator's judgment
12. Treatment with any other investigational agent or participation in another clinical study with therapeutic intent for the lung cancer within 28 days prior to initiating study treatment

Exclusion criteria related to atezolizumab

1. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
2. Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
3. Oral or IV antibiotic treatment. Patients will thus need to have recovered from any infection requiring antibiotics. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
4. Administration of a live, attenuated vaccine within 4 weeks before initiating study treatment or anticipation that such a live attenuated vaccine will be required during the study a) Influenza vaccination is allowed, but should be given during influenza season. However, patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to initiating study treatment, at any time during the study or within 5 months after the last atezolizumab dose.
5. Prior treatment with CD137 agonists or anti-PD-L1 therapeutic antibodies. Patients who have had prior anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) treatment may be enrolled, provided the following requirements are met:

   a) Minimum of 6 weeks from the last dose of anti-CTLA-4 b) No history of severe immune related adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 and 4)
6. Treatment with systemic corticosteroids or other immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents)
7. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Medical Monitor.

   a) The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
8. Patients with history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments done by MRI.
9. Patients not willing to stop treatment with traditional herbal medicines

Exclusion criteria related to radiotherapy

1. Previously irradiated lesions having received the maximum permissible dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 3 months
  Percentage of patients with a complete response or partial response

SECONDARY OUTCOMES:
Overall Survival | 12 months
  Time in months from the first day of study treatment to the date of death
Progression Free-Survival | 12 months
  Time in months from the first day of study treatment until the first evidence of tumour progression

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Martucci, MD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (3):
- Switzerland (3):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Cantonal Hospital of Graubünden (KSGR), Chur
  - Geneva University Hospitals (HUG), Geneva

IPD SHARING:
Plan to Share IPD: No